CLINICAL TRIAL: NCT02379065
Title: Mesh Nebuliser Versus Standard Jet Nebuliser Therapy in Acute Chronic Obstructive Pulmonary Disease in the Emergency Department
Brief Title: Aerogen Nebuliser Versus Standard Nebulised Therapy in Acute Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C&W13/087
Record Dates: First submitted 2015-02-23; First posted 2015-03-04 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control nebuliser treatment (Active Comparator): Both groups will receive the same bronchodilator pharmacotherapy, in keeping with National Institute of Clinical Excellence guidelines. For this arm, nebuliser will be standard of care.
  Interventions:
  Score on the Modified Borg Scale (an interval scale which runs from 0-10, with statements describing level of breathlessness as perceived by the patient) to be completed by both the patient and clinician
  Heart rate (as a measure of severity of exacerbation and an indirect measure of salbutamol dosage)
  Arterial blood gas changes - pH, pO2, pCO2
  Interventions: Device: Phillips Respironic© mask
- Treatment nebuliser treatment (Experimental): Both groups will receive the same bronchodilator pharmacotherapy, in keeping with National Institute of Clinical Excellence guidelines4. For this arm, nebuliser will be Aerogen.
  Interventions:
  Score on the Modified Borg Scale (an interval scale which runs from 0-10, with statements describing level of breathlessness as perceived by the patient) to be completed by both the patient and clinician
  Heart rate (as a measure of severity of exacerbation and an indirect measure of salbutamol dosage)
  Arterial blood gas changes - pH, pO2, pCO2
  Interventions: Device: The Aerogen Aeroneb Solo©

INTERVENTIONS:
Device: The Aerogen Aeroneb Solo©
  Arms: Treatment nebuliser treatment
Device: Phillips Respironic© mask
  Arms: Control nebuliser treatment

SUMMARY:
The investigators are looking at whether a new type of nebuliser (a machine used to deliver drugs to the airways) is better at delivering drugs to the lungs of people with Chronic Obstructive Pulmonary Disease (COPD), compared with the current nebulisers used in Emergency Departments. The investigators will randomly allocate patients who come into the Emergency Department with an acute episode of the COPD into either the standard nebuliser group or the new nebuliser group.

Both groups will receive the same medications, it is only the method of delivering them which will be different.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease presents a significant burden on Emergency Departments and acute medical services, accounting for approximately 90,000 hospital admissions a year, with an average stay lasting 11 days. COPD accounts for 10% of acute hospital admissions, therefore any method of improving health outcomes and reducing the burden on acute services will benefit patients twofold.

Severity of acute COPD is based on clinical indicators such as patient perceived breathlessness, arterial blood gas analysis and respiratory rate. Although breathlessness is a subjective marker, multiple scoring systems have been devised in an attempt to standardise this in order to see an objective improvement in the patient. One of the most commonly used and repeatedly validated scoring systems is the BORG score, which has been shown to effectively demonstrate improvement in breathlessness in the emergency setting .

Nebulised bronchodilator therapy is the mainstay of treatment, as described in the National Institute of Clinical Excellence guidelines. Delivery of bronchodilators (salbutamol and ipratropium) is through a standard facemask - in this Trust it is a Phillips Respironic© mask. Drugs delivery is variable through a nebuliser mask and it is difficult to measure exactly how much of the drug is being delivered to the more distal bronchial tree. Furthermore, this can be highly variable between patients depending on how well the mask fits and patient tolerance, amongst other factors.

Various attempts have been made to improve drug delivery in acute setting such as a spacer and a hood (within paediatric asthmatic patients) , . However, they have all showed that the clinical outcomes are the same regardless of the method of delivery.

Clinical assessment is based on a combination of objective and subjective parameters. Within the Emergency Department, these include both patient and clinician perception of improvement in symptoms (primarily shortness of breath). Assessment also includes more objective measurements such as oxygen saturation, arterial blood gas measurements and end tidal CO2 measurements when available.

There are many challenges that we face specifically within the Emergency Department with patients with COPD. As we are seeing patients as soon as they enter the hospital, initial therapy may have already been administered by the ambulance service so any assessment will be slightly biased and the patient may initially appear better than they actually are. Furthermore, there are often burdens on Emergency Departments during busy periods during the winter, meaning it is not always possible to give patients instant treatment or to be seen immediately by a doctor, particularly if there are more unwell patients based on the triage system.

In addition, some of the more objective measures used in previous trials such as bedside spirometry are not practical in the Emergency Department for several reasons. Firstly, when a patient is acutely short of breath they will not be able to perform spirometry properly. Secondly, as this is not something done routinely in the Emergency Department, both doctors and nurses may not be properly trained to carry this out and we may obtain falsely high or low results.

The Aerogen Aeroneb Solo© is a new nebuliser which is hypothesised to increase drug delivery to peripheral bronchi. Previous studies have showed that it delivers up to 4 times more drug than jet nebulisers and up to 3 times as much as metered dose inhalers. However, this will be its first study with the adapter in human subjects and its first study specifically for COPD.

ELIGIBILITY:
Inclusion Criteria:

* - Documented diagnosis of COPD
* Smoking history of at least 10 pack years (i.e. 20 cigarettes a day for 10 years or equivalent) or other risk factor for COPD in history (e.g. occupational exposure or alpha 1 antitrypsin deficiency)
* Age > 40 years old

Exclusion Criteria:

* - A lack of valid consent from patient (e.g. reduced level of consciousness, dementia)
* Patient unable to speak adequate English - as this study is being conducted in the Emergency Department, there is no access to translators
* Patient refusal
* Ambiguity over diagnosis of COPD e.g. possible underlying asthma
* Patients where an alternate diagnosis (such as congestive cardiac failure) cannot be excluded as the acute medical problem leading to shortness of breath

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Score on the Modified Borg Scale (an interval scale which runs from 0-10, with statements describing level of breathlessness as perceived by the patient) - to be completed by both the patient and clinician | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Roberts, Dr, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom